CLINICAL TRIAL: NCT01837628
Title: Reducing Urethral Pain During Urodynamic Test - Comparison Between Lidocaine Gel and Paraffin Oil
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7/13
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Pain
Keywords: Urodynamic; Paraffin oil; Lidocaine gel; Pain
MeSH Terms: conditions — Pain | interventions — Mineral Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine gel (Active Comparator): Intraurethral Lidocaine gel 2%
  Interventions: Drug: Lidocaine Gel
- Paraffin Oil (Experimental): Intraurethral injection
  Interventions: Drug: Paraffin Oil

INTERVENTIONS:
Drug: Lidocaine Gel
  Arms: Lidocaine gel
Drug: Paraffin Oil
  Arms: Paraffin Oil

SUMMARY:
Our purpose is to compare between intraurethral lidocaine gel and paraffin oil in reducing urethral pain during urodynamic test.

DETAILED DESCRIPTION:
Patients will be randomized into two groups: 1) Lidocaine Gel 2) Paraffin Oil. They will fill out 1 visual analogue scale (0-10) for urethral pain during the test.

ELIGIBILITY:
Inclusion Criteria:

* All men who will be referred for urodynamic test

Exclusion Criteria:

* Active infection
* Permanent Catheter

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue scale (0-10) for pain | up to 1 hour after the procedure
  patients will fill ou the scale before, during and immediately after the test

CONTACTS AND LOCATIONS:
Overall Officials: Kobi Stav, MD, Principal Investigator — Assaf Harofe MC
Locations (1):
- Assaf Harofe Medical Center, Ẕerifin, Israel